CLINICAL TRIAL: NCT01081223
Title: Phase I/II Study To Test The Safety and Efficacy of TVI-Brain-1 As A Treatment For Recurrent Grade IV Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TVAX Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVI-AST-002
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-04

CONDITIONS: Glioma; High Grade Astrocytoma; Glioblastoma Multiforme
Keywords: Brain Neoplasms; Central Nervous System Neoplasms; Brain Diseases; Neoplasms; Nervous System Neoplasms; Glioblastoma; Astrocytoma; Nervous System Diseases; Central Nervous System Diseases; Glioma; Recurrent astrocytoma; Recurrent glioma; Cancer vaccine; Immunotherapy; Killer T cells; Activated T cells; GM-CSF; Low dose IL-2; Activated lymphocytes
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma; Brain Neoplasms; Central Nervous System Neoplasms; Brain Diseases; Neoplasms; Nervous System Neoplasms; Nervous System Diseases; Central Nervous System Diseases | interventions — Cancer Vaccines; Adjuvants, Immunologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TVI-Brain-1 (Experimental): Cancer vaccine plus immune adjuvant Biological/vaccine Other
  Interventions: Biological: Cancer vaccine plus immune adjuvant

INTERVENTIONS:
Biological: Cancer vaccine plus immune adjuvant — Tumor tissue is used for cancer vaccine. Following vaccinations, white blood cells are collected, stimulated and expanded, and are then reinfused. The infusion is followed by a course of low-dose IL-2.

SUMMARY:
TVI-Brain-1 is an experimental treatment that takes advantage of the fact that your body can produce immune cells, called 'killer' white blood cells that have the ability to kill large numbers of the cancer cells that are present in your body. TVI-Brain-1 is designed to generate large numbers of those 'killer' white blood cells and to deliver those cells into your body so that they can kill your cancer cells.

DETAILED DESCRIPTION:
TVI-Brain-1 involves several steps. First, the patient's cancer will be surgically removed to provide cells for the vaccine. Second, the patient will be vaccinated twice with those cells and GM-CSF. Third, the patient's blood will be filtered for white cells which will then be cultured and stimulated to reach a higher (killer) activity level. Fourth, the activated white blood cells will be infused into the patient's bloodstream so that they will be able to attack the cancer. Finally, the entire process starting with vaccination will be repeated, for a total of two rounds of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Informed consent
* Diagnosis of grade IV glioma with progression following standard treatment.
* Must be able to tolerate surgery to provide tumor tissue for vaccine.
* Must be able to produce viable vaccine from tumor tissue.
* Eastern Cooperative Oncology Group (ECOG) performance status must be < 2 or Karnofsky Performance Status must be 70 or greater.
* Negative HIV test.
* Negative for hepatitis B and C virus.
* Respiratory reserve must be reasonable.
* Sufficient renal function.
* Satisfactory blood counts.
* Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Surgically removed cancer reveals that it is not grade IV glioma.
* Concomitant life-threatening disease.
* Active autoimmune disease.
* Currently receiving chemotherapy or biological therapy for the treatment of cancer.
* Currently receiving immunosuppressive drugs for any reason.
* Prior treatment with Avastin or other anti-angiogenesis treatment within 6 months.
* Prior treatment with Gliadel wafers.
* Corticosteroids beyond peri-operative period.
* Psychological, familial, sociological or geographical conditions that do not permit adequate medical follow-up and compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Salacz, M.D., Principal Investigator — St. Luke's Hospital
Locations (1):
- Saint Luke's Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sloan AE, Dansey R, Zamorano L, Barger G, Hamm C, Diaz F, Baynes R, Wood G. Adoptive immunotherapy in patients with recurrent malignant glioma: preliminary results of using autologous whole-tumor vaccine plus granulocyte-macrophage colony-stimulating factor and adoptive transfer of anti-CD3-activated lymphocytes. Neurosurg Focus. 2000 Dec 15;9(6):e9. doi: 10.3171/foc.2000.9.6.10. PMID 16817692
- See also: Sponsor website — http://www.tvaxbiomedical.com

RESULTS

PARTICIPANT FLOW:
Groups:
- TVI-Brain-1: Biological/Vaccine: Cancer vaccine plus immune adjuvant, plus activated white blood cells
Period: Overall Study
Arm/Group | TVI-Brain-1
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11
  Latvia | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing the Incidence of Grade One or Higher Adverse Events
Description: To determine the relative toxicity (safety) of vaccinating recurrent grade IV glioma patients four times with live, attenuated cancer cells combined with granulocyte-macrophage colony-stimulating factor (GM-CSF). Toxicity will be assessed following delivery of each treatment component.
Time Frame: 8 weeks
Population: Number of participants that completed treatment protocol
Measure: Number; unit: participants
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 12
participants | 12

2. Primary Outcome: Immunogenicity as Measured by Delayed Type Hypersensitivity Reactions
Description: The potency of the modified vaccination regimen will be assessed by measuring immune responses following each vaccination. The study is designed to determine whether vaccinating recurrent grade IV glioma subjects four times with attenuated cancer cells stimulates more powerful immune responses than vaccinating subjects twice. Clinical effects also will be measured to determine whether the treatment causes the cancer to regress.
Time Frame: 48 hours
Population: Ten patients developed an immunological response to their tumor as indicated by the delayed type hypersensitivity immune test.
Measure: Count of Participants; unit: Participants
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 12
Participants | 10

3. Secondary Outcome: Overall Survival
Description: Evaluate overall survival of patients
Time Frame: 12 months
Measure: Mean (Full Range); unit: months
Arm/Group | TVI-Brain-1
Number analyzed (Participants) | 12
months | 6.3 [1.8 to 12.6]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Systematic assessments by questionnaires and completion of CRF at each scheduled visit
Arm/Group | TVI-Brain-1
All-Cause Mortality (participants affected / at risk) | 12/12
Serious Adverse Events (participants affected / at risk) | 12/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TVI-Brain-1 (N=12)
coagulopathy (Blood and lymphatic system disorders) | 1 (1)
psychosis postoperative (Psychiatric disorders) | 2 (2)
dehydration (Gastrointestinal disorders) | 1 (1)
asthenia (Nervous system disorders) | 2 (2)
haemorrhage intracranial (Blood and lymphatic system disorders) | 1 (1)
vasogenic cerebral oedema (Injury, poisoning and procedural complications) | 1 (1)
glioblastoma progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12)
weight loss (Investigations) | 1 (1)
hypocalcemia (Investigations) | 3 (3)
hypokalemia (Investigations) | 3 (3)
anxiety (Psychiatric disorders) | 1 (1)
cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TVI-Brain-1 (N=12)
constipation (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 4 (4)
asthenia (Nervous system disorders) | 1 (1)
catheter site inflammation (Skin and subcutaneous tissue disorders) | 1 (1)
fatigue (Nervous system disorders) | 1 (1)
gait disturbance (Nervous system disorders) | 1 (1)
pyrexia (Immune system disorders) | 1 (1)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
gout (Metabolism and nutrition disorders) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1)
anorexia (Gastrointestinal disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 9 (9)
headache (Nervous system disorders) | 4 (4)
hemiparesis (Nervous system disorders) | 1 (1)
hemisensory neglect (Nervous system disorders) | 1 (1)
somnolence (Nervous system disorders) | 1 (1)
vasogenic cerebral edema (Nervous system disorders) | 1 (1)
anxiety (Psychiatric disorders) | 5 (5)
depression (Psychiatric disorders) | 3 (3)
insomnia (Psychiatric disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
small number of participants in study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No